CLINICAL TRIAL: NCT00260832
Title: Randomized Phase 3 Trial of Decitabine Versus Patient's Choice With Physician's Advice of Either Supportive Care or Low-Dose Cytarabine for the Treatment of Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Trial of Decitabine in Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DACO-016
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2011-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Dacogen; Decitabine; Poor or intermediate-risk cytogenetics
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Palliative Care; Decitabine; Single Person

ARMS (2):
- A (Experimental): Subject's choice of treatment with physician's advice. Subjects preselected their preference of supportive care (including IV fluids, nutrition, and antibiotics) or cytarabine. (These represent one intervention.)
  Interventions: Drug: Cytarabine or Supportive Care
- B (Active Comparator)
  Interventions: Drug: Dacogen (decitabine) only

INTERVENTIONS:
Drug: Cytarabine or Supportive Care — Patient's choice with physician's advice of either supportive care (IV fluids, nutrition, and antibiotics as needed) or cytarabine 20 mg/m^2 subcutaneously once daily for the first 10 consecutive days of each 28 day cycle, until progression or unacceptable toxicity develops. (These represent one intervention.)
  Arms: A
Drug: Dacogen (decitabine) only — 20mg/m^2, 1 hour intravenous (IV) for 5 consecutive days of each 28 day cycle. Cycles continue until disease progression or unacceptable toxicity develops.
  Other Names: decitabine
  Arms: B

SUMMARY:
The purpose of this study is to compare the results in older patients who have newly diagnosed or secondary acute myeloid leukemia (AML) and who are to either receive decitabine or patient's choice with the physician's advice of either cytarabine or supportive care medication.

ELIGIBILITY:
Inclusion Criteria:

1. Must have diagnosed acute myeloid leukemia.
2. Must have a life expectancy of at least 12 weeks.
3. Must sign informed consent.

Exclusion Criteria:

1. Must not have acute promyelocytic leukemia (M3 classification)
2. Must not have any other active systemic malignancies.
3. Must not have inaspirable bone marrow.
4. Must not have received previous chemotherapy (except hydroxyurea) for any myeloid disorder.
5. Must not have chronic respiratory disease that requires continuous oxygen use.
6. Must not have received any experimental drug within 4 weeks before randomization.
7. Must not be a candidate for a bone marrow or stem cell transplant within 12 weeks after randomization.
8. Must not have known HIV.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 485 (Actual)
Dates: Start 2005-11; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Global Clinical Development
Locations (108):
- United States (37):
  - Los Angeles, California
  - Fort Myers, Florida
  - Gainesville, Florida
  - Hollywood, Florida
  - Lakeland, Florida
  - Miami, Florida
  - Orange Park, Florida
  - Chicago, Illinois
  - Highland Park, Illinois
  - Terre Haute, Indiana
  - Sioux City, Iowa
  - Wichita, Kansas
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Grosse Pointe Woods, Michigan
  - Kalamazoo, Michigan
  - Neptune City, New Jersey
  - New York, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Sioux Falls, South Dakota
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Galveston, Texas
  - Houston, Texas
  - Temple, Texas
  - Eau Claire, Wisconsin
  - Glendale, Wisconsin
  - Milwaukee, Wisconsin
- Australia (7):
  - Darlinghurst, New South Wales
  - St Leonards, New South Wales
  - South Brisbane, Queensland
  - Adelaide, South Australia
  - East Melbourne, Victoria
  - Parkville, Victoria
  - Perth, Western Australia
- Canada (3):
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Toronto, Ontario
- Croatia (3):
  - Rijeka
  - Zagreb
  - Zalaegerszeg
- Czechia (4):
  - Brno
  - České Budějovice
  - Pilsen
  - Prague
- France (7):
  - Bobigny
  - Créteil
  - Lille
  - Limoges
  - Lyon
  - Nantes
  - Pessac
- Hungary (5):
  - Budapest
  - Győr
  - Gyula
  - Szeged
  - Szombathely
- Mexico City, Mexico
- Poland (7):
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Warsaw
  - Wroclaw
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Târgu Mureş
- Russia (15):
  - Arkhangelsk
  - Astrakhan
  - Barnaul
  - Izhevsk
  - Kirov
  - Kransnodar
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
  - Samara
  - Saratov
  - Tyumen
  - Volgograd
- Serbia (3):
  - Belgrade
  - Niš
  - Novi Sad
- Spain (8):
  - Badalona-Barcelona
  - Barcelona
  - Girona
  - Madrid
  - Palma de Mallorca
  - Pamplona
  - Salamanca
  - Valencia
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Tainan
  - Taipei
- Sutton, United Kingdom

REFERENCES:
- [Derived] Mayer J, Arthur C, Delaunay J, Mazur G, Thomas XG, Wierzbowska A, Ravandi F, Berrak E, Jones M, Li Y, Kantarjian HM. Multivariate and subgroup analyses of a randomized, multinational, phase 3 trial of decitabine vs treatment choice of supportive care or cytarabine in older patients with newly diagnosed acute myeloid leukemia and poor- or intermediate-risk cytogenetics. BMC Cancer. 2014 Feb 6;14:69. doi: 10.1186/1471-2407-14-69. PMID 24498872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 65 centers in 12 countries during the period of 2006 to 2009.
Pre-assignment Details: Prior to randomization, subjects indicated their preference for treatment, with physician's advice, or either cytarabine or supportive care in the event they were randomized to Arm A.
Groups:
- Cytarabine or Supportive Care: Subject's choice of treatment with physician's advice of either supportive care (IV fluids, nutrition, and antibiotics as needed) or cytarabine 20 mg/m^2 given subcutaneously once daily for 10 consecutive days, repeated every 4 weeks. (These represent one intervention.)
- Dacogen (Decitabine) Only: 20 mg/m^2 Dacogen (decitabine) given as 1-hour infusion once daily for 5 consecutive days every 4 weeks.
Period: Overall Study
Arm/Group | Cytarabine or Supportive Care | Dacogen (Decitabine) Only
Started | 243 | 242
Completed | 15 (At study completion, these subjects chose to remain on treatment) | 31 (At study completion, these subjects chose to remain on treatment)
Not Completed | 228 | 211
Not completed — Adverse Event | 26 | 19
Not completed — Progression | 116 | 96
Not completed — Withdrawal by Subject | 15 | 17
Not completed — Physician Decision | 15 | 9
Not completed — Death | 43 | 62
Not completed — Other | 10 | 7
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cytarabine or Supportive Care | Dacogen (Decitabine) Only | Total
Number analyzed (Participants) | 243 | 242 | 485
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.53 (5.67) | 73.14 (5.24) | 73.34 (5.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 105 | 197
  Male | 151 | 137 | 288
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 33 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 213 | 209 | 422
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Patients 65 Years or Older Who Have Newly Diagnosed de Novo or Secondary AML.
Description: The interval from date of randomization to the date of death from any cause or the last date the subject was known to be alive or 5 years whichever occurs first.
Time Frame: The interval from date of randomization to the date of death from any cause or the last date the subject was known to be alive or 5 years whichever occurs first.
Population: The primary population for all efficacy analyses was the Intent-to-treat (ITT) population defined as all subjects randomly allocated to a treatment arm.
Measure: Median (Full Range); unit: months
Arm/Group | Cytarabine or Supportive Care | Dacogen (Decitabine) Only
Number analyzed (Participants) | 243 | 242
months | 5.0 [4.3 to 6.3] | 7.7 [6.2 to 9.2]
Statistical Analysis 1: Comparison: Cytarabine or Supportive Care vs Dacogen (Decitabine) Only; The primary treatment comparison was based on two sided long-rank test stratified by age, cytogenetic risk, ECOG performance status; Test type: Superiority or Other; p = 0.1079, Kaplan-Meier

2. Secondary Outcome: Percentage of Participants With Complete Remission (CR) Plus Complete Remission With Incomplete Platelet Recovery (CRp)
Description: Morphologic CR plus CRp rate where Morphologic leukemia-free state defined as less that (<) 5 percent (%) blasts in an aspirate sample with marrow spicules and a count of greater than or equal to (>=) 200 nucleated cells (there should have been no blasts with Auer rods or persistence of extramedullary disease) plus absolute neutrophil count (ANC) greater than (>)1,000 per microliter (/mcL), platelet count of >=100,000/mcL, and the participant must have been independent of transfusions for at least 1 week before each assessment. There was no duration requirement for confirmation of this designation and Morphologic CR without the requirement of platelet count >=100,000/mcL.
Time Frame: Post randomization when at least one post-baseline bone marrow assessment or peripheral blood count data available (up to 29.5 months)
Population: The primary population for all efficacy analyses was the ITT population defined as all participant randomly allocated to a treatment arm.
Measure: Number; unit: percentage of participants
Arm/Group | Cytarabine or Supportive Care | Dacogen (Decitabine) Only
Number analyzed (Participants) | 243 | 242
percentage of participants | 7.8 | 17.8
Statistical Analysis 1: Comparison: Cytarabine or Supportive Care vs Dacogen (Decitabine) Only; Test type: Superiority; p = 0.0011, Fisher Exact; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.40 to 4.78]

ADVERSE EVENTS:
Arm/Group | Cytarabine or Supportive Care | Dacogen (Decitabine) Only
Serious Adverse Events (participants affected / at risk) | 162/237 | 190/238
Other Adverse Events (participants affected / at risk) | 231/237 | 237/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytarabine or Supportive Care (N=237) | Dacogen (Decitabine) Only (N=238)
Pneumonia (Infections and infestations) | 36 | 48
Sepsis (Infections and infestations) | 10 | 15
Septic Shock (Infections and infestations) | 8 | 15
Bronchopneumonia (Infections and infestations) | 12 | 9
Febrile Neutropenia (Blood and lymphatic system disorders) | 33 | 57
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 21
Anemia (Blood and lymphatic system disorders) | 12 | 15
Neutropenia (Blood and lymphatic system disorders) | 7 | 15
Disease Progression (General disorders) | 31 | 27
Pyrexia (General disorders) | 20 | 23
General Physical Health Deterioration (General disorders) | 14 | 15
Atrial Fibrillation (Cardiac disorders) | 10 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cytarabine or Supportive Care (N=237) | Dacogen (Decitabine) Only (N=238)
Pyrexia (General disorders) | 88 | 114
Disease Progression (General disorders) | 59 | 55
Peripheral Edema (General disorders) | 42 | 50
Pneumonia (Infections and infestations) | 50 | 58
Urinary Tract Infection (Infections and infestations) | 14 | 35
Oral Herpes (Infections and infestations) | 16 | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 86 | 106
Anemia (Blood and lymphatic system disorders) | 73 | 97
Febrile Neutropenia (Blood and lymphatic system disorders) | 54 | 79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No